CLINICAL TRIAL: NCT06613295
Title: Separation Surgery Followed by Stereotactic Ablative Body Radiotherapy Versus Stereotactic Ablative Body Radiotherapy Alone for Spinal Metastases Invading the Spinal Canal: a Randomised, Non-inferiority Trial
Brief Title: Separation Surgery Followed by Stereotactic Ablative Body Radiotherapy (SABR) Versus SABR Alone for Spinal Metastases
Acronym: SABR-MESCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO21003GZA
Record Dates: First submitted 2024-02-06; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor; Spinal Neoplasms; Spinal Tumor
MeSH Terms: conditions — Spinal Neoplasms; Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Separation surgery followed by stereotactic ablative body radiotherapy (Active Comparator): Surgery will take place within 21 days after randomisation. Surgical planning is done by the treating neurosurgeon in the participating center where the patient was included. The goal of separation surgery for intraspinal MESCC is to remove intraspinal epidural disease to allow a margin between the spinal cord (or cauda equina) and the treated radiotherapy volume, and to provide histological diagnosis or confirmation of the metastasis. The decompression should be as minimal invasive as possible, i.e. only intraspinal tumour tissue should be removed, while preserving as much as possible all of surrounding spinal structures. Separation surgery must be followed by SABR after minimum 2 and maximum 4 weeks postoperatively. Image-guided fractionated SABR using a SIB technique to the high-dose PTV will be delivered in 5 fractions of 8 Gy to a total of 40 Gy and to the conventional-dose PTV delivered simultaneously in 5 fractions of 4 Gy to a total of 20 Gy.
  Interventions: Radiation: SABR; Procedure: Separation surgery
- Stereotactic ablative body radiotherapy (Experimental): SABR will start within 21 days of randomisation. Image-guided fractionated SABR using a SIB technique to the high-dose PTV will be delivered in 5 fractions of 8 Gy to a total of 40 Gy and to the conventional-dose PTV delivered simultaneously in 5 fractions of 4 Gy to a total of 20 Gy.
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — SABR
Procedure: Separation surgery — Separation surgery
  Arms: Separation surgery followed by stereotactic ablative body radiotherapy

SUMMARY:
This is a non-inferiority, randomised controlled trial to investigate the effect of stereotactic ablative body radiotherapy (SABR) compared to separation surgery followed by SABR in ambulatory patients with malignant epidural spinal cord compression (MESCC).

The primary objective of the project is investigating the effect of SABR compared to separation surgery followed by SABR in ambulatory patients with MESCC on retaining ambulatory function. The primary endpoint of the study is ambulatory function 3 months post treatment defined as: being able to walk 10m without aid; being able to walk 10m with aid (cane, rollator, one persons help, …); not being able to walk. Secondary outcomes are local control, progression free survival, early and late adverse effects, quality of life, effect on pain and need for reintervention.

The aim is to randomise 128 patients 1:1 to either "separation surgery" followed by SABR (5x 8.0 Gy postoperative) (control arm) vs. SABR alone (5x 8.0 Gy) (study arm).

Patients will be evaluated at 3 and 6 months after treatment with MRI scan, quality of life questionnaires, anamnestic and clinical evaluation at clinical follow ups for assessment of ambulatory function, acute and late toxicity and need for reintervention. Moreover, at 6 weeks, 12 months and 24 months after treatment a teleconsult for assessment of ambulatory function, and need for reintervention will be performed.

DETAILED DESCRIPTION:
In this study, patients with malignant epidural spinal cord compression (MESCC), Bilsky grade 1c, 2 and 3 who are ambulatory with or without aid (rollator, cane, one persons help) will be treated by separation surgery followed by SABR (5x 8.0 Gy postoperative) (control arm) or SABR alone (5x 8.0 Gy) (study arm). The primary objective of the study is investigating the effect of SABR compared to separation surgery followed by SABR in ambulatory patients with MESCC on retaining ambulatory function. The primary endpoint of the study is ambulatory function 3 months post treatment defined as: being able to walk 10m without aid; being able to walk 10m with aid (cane, rollator, one persons help, …); not being able to walk. Secondary outcomes are local control, progression free survival, early and late adverse effects, quality of life, effect on pain and need for reintervention.

For each participant, the study starts once written informed consent is provided and is composed by 4 study phases: a screening phase, randomisation, a treatment phase and a follow-up phase.

The screening phase will allow for assessment of subject eligibility before randomisation and treatment. Demographic data, disease and spinal metastases characteristics and previous anticancer therapies will be recorded. Once all screening procedures are completed, eligibility will be determined according to the inclusion/exclusion criteria. Randomisation will be performed in a 1:1 ratio to the control arm (separation surgery followed by SABR) and the study arm (SABR) using an electronic randomisation tool in the eCRF.

Treatment will be aimed to start as soon as possible, but certainly within 21 days after randomisation (surgery or upfront SABR). Surgical planning is done by the treating neurosurgeon in the participating center where the patient was included. Image-guided fractionated SABR using a SIB technique to the high-dose PTV will be delivered in 5 fractions of 8 Gy to a total of 40 Gy and to the conventional-dose PTV delivered simultaneously in 5 fractions of 4 Gy to a total of 20 Gy.

At 6 weeks (+/-1 week) after the last RT session following information will be obtained (preferentially by digital consult):

1. Ambulatory status defined as: being able to walk 10m without aid, being able to walk 10m with aid (cane, rollator, one persons help, …), not being able to walk
2. WHO performance status
3. Acute and late toxicity assessment: as measured with CTCAE version 5.0
4. Need for re-intervention, date and type of reintervention (surgery or radiotherapy), reason (wound infection, neurologic decline, loss of ability to walk or other)
5. Pain response: VAS pain score
6. Survival data (survival status, date of death, primary cause of death)

At 3 and 6 months (+/-3 weeks) after the last RT session following information will be obtained by physical or digital consult:

1. Ambulatory status defined as: being able to walk 10m without aid, being able to walk 10m with aid (cane, rollator, one persons help, …), not being able to walk
2. WHO performance status
3. Concomitant medications and systemic anticancer therapies
4. QoL according to the EORTC QLQ-C15 & BM22 questionnaires
5. Acute and late toxicity assessment: as measured with CTCAE version 5.0

7. Need for re-intervention, date and type of reintervention (surgery or radiotherapy), reason (wound infection, neurologic decline, loss of ability to walk or other) 6. Pain response: VAS pain score 7. Physical examination: body weight 8. Local control 9. Survival data (survival status, date of death, primary cause of death)

At 12 and 24 months (+/-3 weeks) after the last RT session following information will be obtained (preferentially by digital consult):

1. Ambulatory status defined as: being able to walk 10m without aid, being able to walk 10m with aid (cane, rollator, one persons help, …), not being able to walk
2. Need for re-intervention, type of reintervention
3. Survival data (survival status, date of death, primary cause of death)
4. Local control (only if information is available in medical record as per standard of care)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid malignant tumour (preferentially histologically proven;alternatively obtained by spinal surgical procedure)
* Age 18 years or older
* Histological, radiological or scintigraphical evidence of spinal metastasis (no limitation in the number of sites of metastases)
* Spinal instability neoplastic score (SINS) <13 (i.e. no need for stabilisation of the spine) (see Appendix 6)
* Spinal metastasis with MESCC: ESCC grade 1c, 2 and 3 (see Appendix 7)
* Ambulatory: being able to walk 10m without aid or with aid (cane, rollator, one persons help).
* Life expectancy estimated to be at least 3 months.
* World Health Organization (WHO) Performance Status of 0-2 (some help) (see Appendix 3)
* Patient has given written informed consent.

Exclusion Criteria:

* Contra indication for MRI scan (e.g. pacemaker)
* Previous RT or surgery at the level of the affected vertebrae
* Non-solid primary tumours (e.g. lymphoma, multiple myeloma, germ cell tumours)
* Non ambulatory at presentation
* More than 3 affected vertebrae in one target site
* More than 2 treatment sites
* SINS ≥ 13 (unstable spine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of ambulant patients at 3 months | 3 Months post treatment
  The ambulatory status is scored binary (without or with aid vs not being able to walk)

SECONDARY OUTCOMES:
Local recurrence rate | Up to 24 months post treatment
  Time between date of study registration and date of local recurrence
Time to loss of ambulation | Up to 24 months post treatment
  Time between date of study registration and date of loss of ambulation (in days)
Progression free survival (PFS) | Up to 24 months post treatment
  Time between date of study registration and date of local recurrence
Overall survival | Up to 24 months post treatment
  Time between date of study registration and date of death of any cause or last follow-up
Number of patients with re-intervention and time to re-intervention (surgery, RT, …) | Up to 24 months post treatment
  Time between date of treatment and date of re-intervention
Acute and late toxicity | Up to 6 months post treatment
  Incidence of Adverse Events as assessed by the CTCAE version 5.0
Quality of life measurement by QLQ-BM22 and QLQ-C15-PAL questionnaires | Up to 6 months post treatment
  Difference in QLQ-BM22 and QLQ-C15-PAL scale scores
Pain response (VAS score) | Up to 6 months post treatment
  Improvement by ≥ 2 points on the pain (VAS score) at the treatment site

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Billiet, MD, PhD, Principal Investigator — ZAS Augustinus
Locations (9):
- Belgium (9):
  - OLVZ Aalst, Aalst
  - AZ Klina, Brasschaat
  - UZA, Edegem
  - ZOL, Genk
  - Jessa, Hasselt
  - AZ Groeninge, Kortrijk
  - AZ Sint-Maarten, Mechelen
  - VITAZ, Sint-Niklaas
  - GZA, Wilrijk

IPD SHARING:
Plan to Share IPD: No